CLINICAL TRIAL: NCT03175926
Title: Description of the Ability to Learn How to Handle Inhaler Devices in Asthma - AUDIT
Brief Title: Description of the Ability to Learn How to Handle Inhaler Devices in Asthma
Acronym: AUDIT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Refusal by the ethics committee
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CHUBX 2015/15
Record Dates: First submitted 2017-05-11; First posted 2017-06-05 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Asthma
Keywords: Asthma; inhaler device; handling
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): placebo Diskus® placebo Ellipta® Pulmicort® Turbuhaler®
  Interventions: Device: placebo Diskus®; Device: placebo Ellipta®; Device: Pulmicort® Turbuhaler®
- Group 2 (Experimental): placebo Diskus® placebo Ellipta® Pulmicort® Turbuhaler®
  Interventions: Device: placebo Diskus®; Device: placebo Ellipta®; Device: Pulmicort® Turbuhaler®
- Group 3 (Experimental): placebo Diskus® placebo Ellipta® Pulmicort® Turbuhaler®
  Interventions: Device: placebo Diskus®; Device: placebo Ellipta®; Device: Pulmicort® Turbuhaler®

INTERVENTIONS:
Device: placebo Diskus® — device will be given daily for one week, two puffs per day
Device: placebo Ellipta® — device will be given daily for one week, one puff per day
Device: Pulmicort® Turbuhaler® — device will be given daily for one week, two puffs per day

SUMMARY:
Asthma is a major public health problem. The main treatments against asthma are delivered to the lung through several dry-powder inhaler such as Turbuhaler ®, Diskus® and the new Ellipta® device. In real life, patient's ability to handle a device is not routinely assessed by their practitioner. We hypothesized that many asthmatics cannot properly prepare and prime their device, which may alter the positive effects observed in clinical trials.

DETAILED DESCRIPTION:
The main objective of this study is to describe the handling of inhaler devices (Diskus®, Turbuhaler® and Ellipta®) in patients with asthma.

All participants will use each inhaler device (Diskus®, Turbuhaler® and Ellipta®) daily for one week:

* Two puffs per day (Diskus® and Turbuhaler®),
* One puff per day (Ellipta®). At each visit (day 1, 8, 15 and 22), patients will have a physical exam.

For each inhaler device, 4 video recordings will be performed:

* Video recording #1: Inhalation (one puff) without any instruction of use.
* Video recording #2: Inhalation (one puff) after reading the patient information leaflet.
* Video recording #3: Inhalation (one puff) after watching a standardized video demonstrating correct inhaler technique.
* Video recording #4: inhalation (one puff) after seven days of daily use. The patient will be asked to fulfill a satisfaction survey about each inhaler device.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged more than 18 years
* Written informed consent
* Diagnosis of asthma according to international guidelines (GINA 2017)
* Social security or health insurance
* Women using an effective method of birth control.

Exclusion Criteria:

* Previous treatment with Ellipta®, Diskus® or Turbuhaler®
* Asthma exacerbation within 6 weeks before inclusion
* Subject having close contacts with devices (Ellipta®, Diskus® or Turbuhaler®) users, currently or in the past
* Severe asthma
* Hypersensitivity to budesonide
* Chronic psychiatric disease
* Medical condition that may affect handling of inhaler devices
* Subject deprived of his/her liberty
* Protected adult
* Subject in exclusion period related to another protocol
* Pregnant or breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-12-01 (Estimated); Primary Completion 2018-09-01 (Estimated); Study Completion 2018-09-01 (Estimated)

PRIMARY OUTCOMES:
Critical errors | Day 8 of each treatment
  Assessment of the presence of at least a critical error in the use of the inhalation system, from standardized checklist

SECONDARY OUTCOMES:
Non device-dependent errors | Day 8 of each treatment
  Assessment of the presence of non device-dependent errors from standardized checklist with first device
Time for drug administration | Day 8 of each treatment
  Measure of the necessary time for drug administration with each device
Patient satisfaction questionnaire | Day 8 of each treatment
  Questionnaire of satisfaction about the use of each device

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Olivier GIRODET, MD, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- Bordeaux University Hospital, Bordeaux, France

IPD SHARING:
Plan to Share IPD: Undecided